CLINICAL TRIAL: NCT03670420
Title: The Application of Honey on Perineal Sutures: a Randomized Controlled Clinical Trial
Brief Title: The Application of Honey on Perineal Sutures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marie-Julia GUITTIER, Associate Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00995
Record Dates: First submitted 2018-09-04; First posted 2018-09-13 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Perineal Tear; Pain; Burns
MeSH Terms: conditions — Pain; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical honey in addition to standard care (Experimental): In addition to the usual care provided by the maternity unit, women allocated to this group apply honey on first and second degree perineal tears, episiotomies and anterior vulvar tears twice a day for four days from randomization.
  Interventions: Other: Medical honey
- Standard care (No Intervention): This group benefits from the standard care offered by the maternity: hygiene advice, analgesics, ice packs, buoys and positioning.

INTERVENTIONS:
Other: Medical honey — The investigators use Medihoney®, a medical honey released by the DermaSciences.
  Arms: Medical honey in addition to standard care

SUMMARY:
Evaluate the effect of honey on perineal tears or episiotomies pain associated or not with anterior vulvar tears after vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

* Major women
* Giving birth vaginally in the maternity of Geneva university hospital
* First and second degree perineal tears or episiotomy
* French speaking women
* The day of the delivery

Exclusion Criteria:

* Allergic to honey and bees
* Drug use
* postpartum hemorrhage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Mean change between groups in perceived pain scores on the visual analog scale at day 1 post-partum | Day 1
  A Visual Analogue Scale (VAS) is used by women to evaluate perceived pain. The score is determined by measuring the distance (mm) on the 100 mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0 to 100 mm. A higher score indicates greater pain intensity.
  Pain is evaluate at two different times (day 1 and 4) in order to objectify changes between the two groups and at the two measurement times.
Saint Antoine questionnaire to measure perceived pain at day 1 post-partum | Day 1
  Participants complete the Saint Antoine questionnaire (1), a french version of the short form Mcgill pain questionnaire. Mcgill pain questionnaire can be used to evaluate a person experiencing significant pain. Women use a Likert 5 points scale to assess words that describe their pain : Absent, Low, Moderate, High Extremely, High.
  Pain is evaluate at two different times (day 1 and 4) in order to objectify changes between the two groups and at the two measurement times.
Mean change between groups in perceived pain scores on the visual analog scale at day 4 post-partum | Day 4
  A Visual Analogue Scale (VAS) is used by women to evaluate perceived pain. The score is determined by measuring the distance (mm) on the 100 mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0 to 100 mm. A higher score indicates greater pain intensity.
  Pain is evaluate at two different times (day 1 and 4) in order to objectify changes between the two groups and at the two measurement times.
Saint Antoine questionnaire to measure perceived pain at day 4 post-partum | Day 4
  Participants complete the Saint Antoine questionnaire (1), a french version of the short form Mcgill pain questionnaire. Mcgill pain questionnaire can be used to evaluate a person experiencing significant pain. Women use a Likert 5 points scale to assess words that describe their pain : Absent, Low, Moderate, High Extremely, High.
  Pain is evaluate at two different times (day 1 and 4) in order to objectify changes between the two groups and at the two measurement times.

SECONDARY OUTCOMES:
Mean change between groups in peceived burn scores on the visual analog scale at day 1 post-partum | Day 1
  A Visual Analogue Scale (VAS) is used to measure burning sentation. The score is determined by measuring the distance (mm) on the 100 mm line between the "no burn" anchor and the patient's mark, providing a range of scores from 0 to 100 mm. A higher score indicates greater burn intensity.
  Burning sensation is evaluate at two different times (day 1 and 4) in order to objectify changes between the two groups and at the two measurement times.
Proportions between groups in a Likert scale to measure women satisfaction about honey application on perineal sutures at day 1 | Day 1
  Women included in the intervention group complete a five points Likert scale ( Not at all, Very few, Few, Satisfied, Very satisfied) to evaluate their satisfaction with the application of honey on their perineal sutures.
  Woman satisfaction about honey application is evaluate at two different times (day 1 and 4) in order to objectify changes between the two measurement times.
Mean change between groups in peceived burn scores on the visual analog scale at day 4 post-partum | Day 4
  A Visual Analogue Scale (VAS) is used to measure burning sentation. The score is determined by measuring the distance (mm) on the 100 mm line between the "no burn" anchor and the patient's mark, providing a range of scores from 0 to 100 mm. A higher score indicates greater burn intensity.
  Burning sensation is evaluate at two different times (day 1 and 4) in order to objectify changes between the two groups and at the two measurement times.
Proportions between groups in a Likert scale to measure women satisfaction about honey application on perineal sutures at day 1 | Day 4
  Women included in the intervention group complete a five points Likert scale ( Not at all, Very few, Few, Satisfied, Very satisfied) to evaluate their satisfaction with the application of honey on their perineal sutures.
  Woman satisfaction about honey application is evaluate at two different times (day 1 and 4) in order to objectify changes between the two measurement times.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] https://doi.org/10.1007/s11724-008-0083-6
- See also: The psychometric caractéristiques of the Saint Antoine Questionnaire — https://doi.org/10.1007/s11724-008-0083-6